CLINICAL TRIAL: NCT01497470
Title: An Open-Label, One-Arm, One-Sequence Crossover Drug-Drug Interaction Study in Advanced Solid Tumor Subjects Subjects to Evaluate the Potential Effect of Custirsen (OGX-011) on the Pharmacokinetics of Paclitaxel
Brief Title: A Clinical Study in Cancer Patients to Investigate the Potential Impact of Custirsen, on the Blood Levels of the Chemotherapeutic Drug, Paclitaxel, When Given Together as Part of a Treatment Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TV1011-DDI-105
Record Dates: First submitted 2011-12-09; First posted 2011-12-22 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: paclitaxel; carboplatin; custirsen; drug-drug interaction; pharmacokinetics; cancer
MeSH Terms: conditions — Neoplasms | interventions — OGX-011; Paclitaxel; Carboplatin

ARMS (1):
- Paclitaxel/carboplatin with custirsen (Experimental): Custirsen added to standard paclitaxel/carboplatin chemotherapy
  Interventions: Drug: Custirsen, paclitaxel and carboplatin

INTERVENTIONS:
Drug: Custirsen, paclitaxel and carboplatin — Custirsen (640 mg IV over 2 hours) will be administered weekly on Days 1, 8, and 15 of each 21 day cycle. Paclitaxel (200 mg/m2 IV over 3 hours) and carboplatin (AUC 6.0 mg/mL/min IV over 30 minutes) will be administered on Day 1 of each 21 day cycle

SUMMARY:
The primary goal of this study is to determine if custirsen has an effect on the way the body distributes and gets rid of paclitaxel, the standard administered chemotherapy. The study will also evaluate if custirsen influences the way the body distributes and gets rid of carboplatin (another standard administered chemotherapy) and will measure custirsen blood levels in this cancer population. Finally, the study will evaluate the safety and tolerability of adding custirsen to the standard paclitaxel/carboplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a solid tumor that is refractory to standard therapies and is not amenable to treatment with established curative or palliative therapies and for whom paclitaxel and carboplatin is deemed an acceptable treatment by the investigator
* Males or females ≥18 years of age
* Life expectancy of ≥12 weeks
* Minimum of 1 lesion
* ECOG performance status of 0, 1 or 2
* Adequate bone marrow reserve
* Adequate renal and liver function

Exclusion Criteria:

* Brain metastases that are symptomatic or require ongoing treatment
* Major trauma or surgery within last 2 months, acute infection within 2 weeks (14 days), or radiotherapy, chemotherapy, immunotherapy or hormonal therapy within past 4 weeks
* Persistent grade 2 or greater toxicity related to prior therapy
* Grade 2 or greater peripheral neuropathy
* Recent or current use of Cyp3A4, Cyp2C8 or P-gp inhibitors
* Recent or current use of CYP enzyme inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of custirsen on paclitaxel pharmacokinetics | 0, 1, 2, 3, 3.25, 3.67, 4.5, 6, 8, 12, 24 and 48 hours after the start of paclitaxel infusion
  The maximum peak concentration of paclitaxel after administration.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of adding custirsen to standard paclitaxel/carboplatin chemotherapy | 0, 1, 2, 3, 3.25, 3.67, 4.5, 6, 8, 12, 24 and 48 hours after the start of paclitaxel infusion

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Teva Investigational Site 002, Detroit, Michigan
  - Teva Investigational Site 001, Dallas, Texas
  - Teva Investigational Site 003, San Antonio, Texas
  - Teva Investigational Site 004, Tacoma, Washington